CLINICAL TRIAL: NCT00118157
Title: A Phase II Study of GW572016 and Tamoxifen in Patients With Metastatic Breast Cancer Resistant to Single-Agent Tamoxifen
Brief Title: Lapatinib and Tamoxifen in Treating Patients With Locally Advanced or Metastatic Breast Cancer That Did Not Respond to Previous Tamoxifen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00080; NCI-2009-00080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000433388; C-2876 (Other: Wayne State University/Karmanos Cancer Institute); 6724 (Other: CTEP); P30CA022453 (NIH); U01CA062487 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Estrogen Receptor Positive; Male Breast Carcinoma; Progesterone Receptor Positive; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Lapatinib; Tamoxifen

ARMS (1):
- Treatment (lapatinib, tamoxifen) (Experimental): Patients receive lapatinib ditosylate PO daily and tamoxifen citrate PO daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lapatinib Ditosylate; Drug: Tamoxifen Citrate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lapatinib Ditosylate — Given PO
  Other Names: Tykerb
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI-46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide

SUMMARY:
This phase II trial studies how well giving lapatinib ditosylate together with tamoxifen citrate works in treating patients with breast cancer that has spread from where it started to nearby tissue or lymph nodes or to other areas of the body and did not respond to previous treatment with tamoxifen citrate. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen citrate may fight breast cancer by blocking the use of estrogen by the tumor cells. Sometimes when tamoxifen citrate is given, it does not stop the growth of tumor cells. The tumor is said to be resistant to tamoxifen citrate. Giving lapatinib ditosylate together with tamoxifen citrate may reduce drug resistance and allow the tumor cells to be killed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (complete response and partial response) of tamoxifen (tamoxifen citrate) and GW572016 (lapatinib ditosylate) in women with hormone refractory, metastatic breast cancer.

II. To describe the changes in phosphorylation of epidermal growth factor receptor (EGFR), human EGFR 2 (her2), protein B kinase (AKT) kinase, mitogen activated protein kinase (MAPK), estrogen receptor (ER)-Serine (Ser) 118, and ER-Ser167 in tumor tissue after administration of tamoxifen and GW572016.

OUTLINE:

Patients receive lapatinib ditosylate orally (PO) daily and tamoxifen citrate PO daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Primary adenocarcinoma of the breast confirmed by histology or cytology
* Locally advanced or metastatic disease not amenable to surgery or radiation therapy with curative intent
* Estrogen and/or progesterone receptor positive cancer
* Patients have failed hormonal manipulation with tamoxifen, either showing no response (primary resistance) to initial therapy or relapse/progression after showing initial response (secondary failure)
* At least 1 measurable (target) lesion (i.e. any malignant tumor mass that can be accurately measured in at least 1 dimension, >= 20 mm with conventional radiographic techniques or >= 10 mm with magnetic resonance imaging [MRI] or spiral computerized tomography [CT] scans), in a previously un-irradiated area
* No more than 450 mg/m^2 of prior doxorubicin
* Life expectancy >= 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Creatinine (Cr) =< upper limit of normal (ULN) or Cr clearance > 60 mL/min/m^2
* Total bilirubin =< 1.5 x ULN
* Alanine aminotransferase (ALT) =< 1.5 x ULN or =< 3 x ULN with liver metastases
* Aspartate aminotransferase (AST) =< 5 x ULN or =< 3 x ULN with liver metastases
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or multi gated acquisition scan (MUGA) scan; (note that baseline and on-treatment scans should be performed using the same modality and preferably at the same institution)
* Patients on oral anticoagulants (Coumadin, warfarin) should either be switched to low molecular weight heparin or have a very close monitoring of international normalized ratio (INR), if continued on Coumadin
* Negative serum pregnancy test within 7 days of enrollment for pre-menopausal women and women within 6 months of menopause; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; both men and women should be counseled in contraceptive use due to unknown effects of the drug on the fetus and breast feeding should be avoided
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow and retain oral medication

Exclusion Criteria:

* Patients who have had prior treatment with EGFR and or Her-2 targeting therapies (prior trastuzumab combined with chemotherapy in the adjuvant setting only is allowed, but the combination of trastuzumab with hormonal therapy is not allowed)
* Current treatment with any other anti-neoplastic agent, including trastuzumab; patients may continue to receive zoledronic acid for bone metastases or hypercalcemia
* Radiation therapy within 2 weeks of enrollment or surgery within 4 weeks
* Rapidly progressive disease in major organs (i.e. lymphangitic spread, bulky liver metastasis) or known brain/leptomeningeal metastatic disease requiring active therapy; (patients with asymptomatic, stable previously treated metastases to the central nervous system and surrounding tissues are eligible; however patients must not have a requirement for corticosteroids due to central nervous system metastases at the time of study entry)
* Any of the following conditions within 6 months of enrollment: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, coronary/peripheral artery bypass grafting; patients who have experienced a pulmonary embolus, deep venous thrombosis or other clinically significant thromboembolic event within 6 months of enrollment are eligible if they are clinically stable on anticoagulation therapy
* Pregnancy or breast feeding; breastfeeding should be discontinued if the mother is treated with GW572016; female patients must agree to use effective contraception during the study period, be surgically sterile, or be post-menopausal; in addition, male patients will be required to use effective contraception during the study period or be surgically sterile; the definition of effective contraception will be based on the judgment of the investigator
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016
* Patients with gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Treatment with any agents that interact with cytochrome P450 3A should be avoided and used with caution, if necessary; when possible, patients should be switched to alternative medications; patients requiring anticoagulation should either be switched to a low molecular weight heparin injection or have a very close monitoring of INR, if continued on Coumadin
* Previous (within 5 years of enrollment) or current malignancies at other sites, except adequately treated basal cell or squamous cell skin cancers and carcinoma in situ of the cervix
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-05; Primary Completion 2011-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaina Gartner, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Harper University Hospital - DMC, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Patients receive oral lapatinib and oral tamoxifen once daily on days 1-28.
  lapatinib ditosylate: Given orally
  tamoxifen citrate: Given orally
Period: Overall Study
Arm/Group | Arm 1
Started | 19
Completed | 7
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — Death | 8
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 57 [32 to 84]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (Complete and Partial) Assessed by Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Arm 1
Number analyzed (Participants) | 17
participants | 1 [1 to 27]

2. Secondary Outcome: Changes in Phosphorylation in Tumor Tissue of Epidermal Growth Factor Receptor (EGFR), HER2, AKT Kinase, MAPK, ER-Ser118, and ER-SER167
Time Frame: Baseline and at 21 days
Population: Data were not collected due to feasibility.
Arm/Group | Treatment (Lapatinib, Tamoxifen)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 19/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=19)
Hemolysis (Blood and lymphatic system disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 19 (19)
Death NOS (General disorders) | 10 (10)
Fatigue (General disorders) | 13 (13)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 4 (4)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
White blood cell decreased (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=19)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 4 (4)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Weight loss (Investigations) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gait disturbance (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitation in this study was poor enrollment. The small number of cases makes the interpretation of results difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less